CLINICAL TRIAL: NCT03485534
Title: Evaluate the Efficacy and Safety of Switching to Tenofovir Disoproxil From Tenofovir Disoproxil Fumarate in Chronic Hepatitis B Patients Who Pretreated With Tenofovir Disoproxil Fumarate
Brief Title: Evaluate the Efficacy and Safety to Tenofovir Disoproxil in Chronic Hepatitis B Patients
Acronym: HBV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Collaborators: C&R Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DW_TEN001
Record Dates: First submitted 2018-03-27; First posted 2018-04-02 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, Parallel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenofovir Disoproxil (Experimental): Tenofovir Disoproxil 245mg, a daily dose for 48 weeks
  Interventions: Drug: Tenofovir Disoproxil
- Tenofovir Disoproxil Fumarate (Placebo Comparator): Tenofovir Disoproxil Fumarate 300mg, a daily dose for 48 weeks
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — Viread 300mg
  Other Names: Viread
  Arms: Tenofovir Disoproxil Fumarate
Drug: Tenofovir Disoproxil — Virehepa 245mg
  Other Names: Virehepa
  Arms: Tenofovir Disoproxil

SUMMARY:
This study evaluates the efficacy and safety of switching to Tenofovir Disoproxil from Tenofovir Disoproxil Fumarate in Chronic Hepatitis B Patients who pretreated with Tenofovir Disoproxil Fumarate.

In Open-Label, phase 3 studies, we randomly assigned patients with hepatitis B e antigen (HBeAg)-negative or HBeAg-positive chronic HBV infection to receive Tenofovir Disoproxil or Tenofovir Disoproxil Fumarate (ratio, 2:1) once daily for 48 weeks

DETAILED DESCRIPTION:
Tenofovir Disoproxil and Tenofovir Disoproxil Fumarate is a nucleotide analogue and a potent inhibitor of human immunodeficiency virus type 1 reverse transcriptase and hepatitis B virus (HBV) polymerase.

The primary efficacy end point at week 48 of this study was defined as the combination of an HBV DNA level of less than 400 copies per milliliter and histologic improvement .

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B virus (HBV) infection, defined as positive serum hepatitis B s-antigen (HBsAg) for at least 6 months.
* HBeAg negative and HBeAb positive at screening

Exclusion Criteria:

* Pregnant women, women who are breast feeding, or women who believe they may wish to become pregnant during the course of the study
* Males and females of reproductive potential who are unwilling to use an effective method of contraception during the study.
* Decompensated liver disease defined as conjugated bilirubin > 1.5 x ULN, prothrombin time (PT) > 1.5 x ULN, platelets < 75,000/mL, serum albumin < 3.0 g/dL, or prior history of clinical hepatic decompensation (eg, ascites, jaundice, encephalopathy, variceal hemorrhage)
* Significant renal, cardiovascular, pulmonary, or neurological disease
* currently receiving therapy with immunomodulators (eg, corticosteroids, etc.), investigational agents, nephrotoxic agents, or agents susceptible of modifying renal excretion

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
HBV DNA inhibition | 48weeks
  plasma HBV DNA level of less than 400 copies per milliliter

SECONDARY OUTCOMES:
viral suppression | 24weeks
  an HBV DNA level of <400 copies per milliliter

CONTACTS AND LOCATIONS:
Overall Officials: Youngsuk Lim, PHD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided